CLINICAL TRIAL: NCT02822729
Title: A Long-term Open-label Study of DE-117 Ophthalmic Solution Monotherapy and Concomitant Use of DE-117 Ophthalmic Solution With Timolol Ophthalmic Solution in Patients With Open-angle Glaucoma or Ocular Hypertension : RENGE Study
Brief Title: A Long-term Study of DE-117 Ophthalmic Solution Monotherapy and Concomitant Use of DE-117 Ophthalmic Solution With Timolol Ophthalmic Solution in Patients With OAG or OH: RENGE Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01171504
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Open Angle Glaucoma or Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DE-117 ophthalmic solution (Group1) (Experimental): Monotherapy
  Interventions: Drug: DE-117 ophthalmic solution
- DE-117 ophthalmic solution (Group2) (Experimental): Monotherapy
  Interventions: Drug: DE-117 ophthalmic solution
- DE-117 ophthalmic solution + Timolol (Group3) (Other): Concomitant Use
  Interventions: Drug: DE-117 ophthalmic solution; Drug: Timolol ophthalmic solution

INTERVENTIONS:
Drug: DE-117 ophthalmic solution
Drug: Timolol ophthalmic solution
  Arms: DE-117 ophthalmic solution + Timolol (Group3)

SUMMARY:
The purposes of this study are to evaluate the long-term safety and intraocular pressure-lowering efficacy of DE-117 ophthalmic solution monotherapy and concomitant use of DE-117 ophthalmic solution with timolol ophthalmic solution 0.5% in patients with open angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with open angle glaucoma or ocular hypertension

Exclusion Criteria:

* Patients at risk of progression of visual field loss
* Patients with severe visual field defect
* Patients with any diseases that preclude participation in this study for safety reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of adverse events | Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Derived] Aihara M, Lu F, Kawata H, Iwata A, Odani-Kawabata N. Twelve-month efficacy and safety of omidenepag isopropyl, a selective EP2 agonist, in open-angle glaucoma and ocular hypertension: the RENGE study. Jpn J Ophthalmol. 2021 Nov;65(6):810-819. doi: 10.1007/s10384-021-00868-y. Epub 2021 Sep 8. PMID 34495425